CLINICAL TRIAL: NCT03676491
Title: Music to Improve Sleep Quality in Adults With Depression and Insomnia: a Randomized Controlled Trial Using Mixed Methods
Brief Title: Music to Improve Sleep Quality in Adults With Depression and Insomnia
Acronym: MUSTAFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Health Research Foundation (Other); The Obel Family Foundation (Unknown); Aase & Ejnar Danielsens Foundation (Unknown)
Responsible Party: Principal Investigator, Helle Nystrup Lund, Music Therapist, Ph.d. student, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20170055; N-20170055 (Registry Identifier: 296056)
Record Dates: First submitted 2018-08-29; First posted 2018-09-18 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Insomnia; Depression
Keywords: music; depression; sleep disturbances; insomnia; quality of life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Parasomnias

STUDY DESIGN:
Intervention Model Description: The study design is an explanatory mixed methods design in two parts. The first part is a two-arm parallel group, single center randomized controlled trial (n=120). Experimental group and waitlist control group receive standard treatment according to national guidelines. The experimental group use a sound pillow and The Music Star App at bedtime as a sleep aid in 4 weeks.The second part is an interview study (n=4). Qualitative data from a semi-structured interview on the use of music and sleep are used to discuss findings from the RCT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Music Intervention: Participants listen to music minimum 30 minutes at bedtime for a period of 4 weeks wearing accelerometer.
  Participants are monitored for a 4 week follow up period wearing accelerometer
  Interventions: Other: Music Intervention
- Waitlist Control Group (No Intervention): No intervention: Participants are monitored for a period of 4 weeks wearing accelerometer.
  Participants are monitored for a 4 week follow up period wearing accelerometer.

INTERVENTIONS:
Other: Music Intervention — Music intervention
  Arms: Experimental Group

SUMMARY:
Insomnia is a common sleep disorder for patients with depression. This has a major impact on the quality of life for the individual.

The aim is to investigate, whether music intervention is effective in

1. improving sleep quality,
2. reducing symptoms of depression and
3. improving quality of life

Participants use a sound pillow and selected music in the The Music Star app at home as a sleep aid in 4 weeks.

DETAILED DESCRIPTION:
Depression is a common health problem in Denmark with a prevalence for depression of 17-18%. Depression has serious personal and social consequence. Sleep disorders are common in patients with depression. Resolving sleep disturbances in depression may prevent worsening of symptoms and relapse.

Music listening is widely used as a sleep aid. A study from the Cochrane library shows consensus that music may be helpful to improve sleep quality in insomnia. It remains unclear if music listening is helpful to patients with depression as it is to a broader population.

A randomized controlled trial address the use of music as a supplementary treatment to improve sleep in depression.

ELIGIBILITY:
Inclusion Criteria:

* Out patients in treatment for depression in psychiatry, Unit for Depression, Aalborg University Hospital.
* ICD-10 diagnosis of unipolar depression F32 or F33.
* Sleeping problems identified by HAM-D by a total score of 3 on sleep items 4-6, or a single score = 2 on at least one sleep item.
* Following treatment standards according to national guidelines.(pharmacological treatment, psychotherapy, psycho education, Electro Convulsive Therapy).
* 4 weeks of treatment and/or in stabilized pharmacological treatment

Exclusion Criteria:

* ICD-10 diagnosis of depression F32 or F33 and psychotic episodes
* substance or alcohol abuse
* sentence to treatment by law
* restless legs syndrome
* obstructive sleep apnoea or other organic sleep disorders
* hearing loss
* dislike of music

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Sleep Quality - subjective | Change of sleep quality from baseline at 4 weeks
  Questionnaire PSQI-DK on self reported sleep measuring subjective sleep quality, sleep latency, sleep duration, sleep disturbances, daytime dysfunctions and use of antidepressant agents

SECONDARY OUTCOMES:
Sleep Quality - subjective | Change of sleep quality from baseline at 8 weeks
  Questionnaire PSQI-DK on self reported sleep measuring subjective sleep quality, sleep latency, sleep duration, sleep disturbances, daytime dysfunctions and use of antidepressant agents.
Sleep Quality - objective | Change of sleep quality from baseline at 4 weeks
  Accelerometer Axivity Ax3 data logger carried as a hand wrist bracelet at night. A sleep analysis function by a generic algorithm provide data on sleep estimates.
Sleep Quality - objective | Change of sleep quality from baseline at 8 weeks
  Accelerometer Axivity Ax3 data logger carried as a hand wrist bracelet at night. A sleep analysis function by a generic algorithm provide data on sleep estimates.
Symptoms of depression | Change of depression level from baseline at 4 weeks
  The Hamilton Depression Rating Scale (HAM-D17). The scale consist of 17 items. Total score range is 0-52. Higher numbers represent more severe symptoms.
Symptoms of depression | Change of depression level from baseline at 8 weeks
  The Hamilton Depression Rating Scale (HAM-D17). The scale consist of 17 items. Total score range is 0-52. Higher numbers represent more severe symptoms.
Quality of life measuring subjective well-being | Change of quality of life from baseline at 4 weeks
  The World Health Well-Being Index (WHO-5)
Quality of life measuring subjective well-being | Change of quality of life from baseline at 8 weeks
  The World Health Well-Being Index (WHO-5)
Quality of life measuring subjective psychological health, physical health, social relationships and environment. | Change of quality of life from baseline at 4 weeks
  The World Health Organization Quality of Life (WHOQOL-Bref)
Quality of life measuring subjective psychological health, physical health, social relationships and environment. | Change of quality of life from baseline at 8 weeks
  The World Health Organization Quality of Life (WHOQOL-Bref)

OTHER OUTCOMES:
Duration of music intervention | 4 week music intervention period
  log file data on duration of music intervention

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Risom Kristensen, Professor, Study Director — Aalborg University, Doctoral School in Medicine, biomedical science and technology
Locations (1):
- Unit for Depression, Psychiatry, Aalborg, Denmark

REFERENCES:
- [Background] Fava M. Daytime sleepiness and insomnia as correlates of depression. J Clin Psychiatry. 2004;65 Suppl 16:27-32. PMID 15575802
- [Background] Jespersen KV, Koenig J, Jennum P, Vuust P. Music for insomnia in adults. Cochrane Database Syst Rev. 2015 Aug 13;2015(8):CD010459. doi: 10.1002/14651858.CD010459.pub2. PMID 26270746
- [Derived] Jespersen KV, Pando-Naude V, Koenig J, Jennum P, Vuust P. Listening to music for insomnia in adults. Cochrane Database Syst Rev. 2022 Aug 24;8(8):CD010459. doi: 10.1002/14651858.CD010459.pub3. PMID 36000763
- [Derived] Lund HN, Pedersen IN, Heymann-Szlachcinska AM, Tuszewska M, Bizik G, Larsen JI, Drago A, Kulhay E, Larsen A, Sorensen HO, Gronbech B, Bertelsen LR, Valentin JB, Mainz J, Johnsen SP. Music to improve sleep quality in adults with depression-related insomnia (MUSTAFI): randomized controlled trial. Nord J Psychiatry. 2023 Feb;77(2):188-197. doi: 10.1080/08039488.2022.2080254. Epub 2022 Jun 13. PMID 35697087
- [Derived] Lund HN, Pedersen IN, Johnsen SP, Heymann-Szlachcinska AM, Tuszewska M, Bizik G, Larsen JI, Kulhay E, Larsen A, Gronbech B, Ostermark H, Borup H, Valentin JB, Mainz J. Music to improve sleep quality in adults with depression-related insomnia (MUSTAFI): study protocol for a randomized controlled trial. Trials. 2020 Apr 3;21(1):305. doi: 10.1186/s13063-020-04247-9. PMID 32245512